

# **Clinical Study Protocol:**

### Patient-Assisted Compression – Impact on Image Quality and Workflow

(124.03-2017-GES-0002)

Version: 1.0; 22/May/2017

**Sponsor:** General Electric Company, acting through its GE Healthcare Business

3000 N. Grandview Blvd Waukesha, WI 53188

**Sponsor Contact:** Sara Lam, Clinical Affairs Project Manager

*Tel*: 1-262-548-2369

E-mail: Sara.J.Lam@ge.com

**Medical Monitor:** Ron von Jako, MD, PhD, Medical Director

*Tel*: 1-617-669-3200

E-mail: Ron.VonJako@med.ge.com

Investigational Product: Patient-Assisted Compression, Senographe Pristina Modality: Imaging,

Women's Health

# FOR QUALIFIED INVESTIGATORS, STUDY STAFF, AND THEIR ETHICS COMMITTEE(S) ONLY

#### **CONFIDENTIALITY STATEMENT**

Information in this RESEARCH STUDY PROTOCOL is for investigators, site personnel involved with the study, ethics committee(s), and/or their authorized representative(s) except as required to obtain consent from study participants or as otherwise required by law. Once signed, the terms of the protocol are binding for all parties.

 GE MWS DOC1991348 Ver: 1.0; 22/May/2017 **Study Title:** Patient-Assisted Compression – Impact on Image Quality and Workflow **Study No:** 124.03-2017-GES-0002



The Sponsor and Investigator have approved this protocol version, and I confirm hereby to conduct the study according to the protocol and in accordance with applicable principles of the World Medical Association Declaration of Helsinki and Good Clinical Practice (GCP) guidelines as per ISO 14155:2011, any conditions of approval imposed by the reviewing EC or governing regulatory body, and applicable laws and regulations. The investigator should not deviate from this protocol except for emergency use. I have read and understood and agree to abide by all the conditions and instructions contained in this protocol.

Mully Mally Date

Investigator Signature

Print Name

BRRH WOMEN'S INSTRATE 690 MEADOWS RO. BOLARATON SE 33486

Site Name, Department, Address

Principal Investigator at study site:



# **Table of Contents**

| | nent and Version Control | |
|---|---|---|
| List of | Abbreviations and Terms | 6 |
| | Synopsis | |
| Admin | istrative Structure of Investigation | 11 |
| 1. Ba | ckground and Justification | 12 |
| 1.1 | Screening Mammography and Patient-Assisted Compression | 12 |
| 1.2 | Controls and Minimization of Bias | 12 |
| 2. De | vice/Product Description | |
| 2.1 | Identity, Mechanism, and Function of Investigational Device | |
| 2.2 | Mammography Review Workstation | |
| 2.3 | Intended Use | |
| 2.4 | Comparator | |
| 2.5 | Concomitant/Ancillary Administrations | |
| 2.6 | Accountability | |
| 2.7 | Anticipated Risks and Benefits | |
| | udy Objectives and Endpoints | |
| 3.1 | Purpose of the Study | |
| 3.2 | Study Endpoints | |
| 3.3 | Summary of Study Design | |
| | udy Design | |
| 4.1 | Study Population | |
| 4.2 | Number Subjects<br>Protection of Vulnerable Subjects | |
| 4.3<br>4.4 | Eligibility Criteria | |
| 4.4<br>4.5 | Recruiting and Screening | |
| 4.5<br>4.6 | Breast of Interest Randomization | |
| 4.7 | Criteria for Withdrawal/Discontinuation | |
| | udy Procedures | |
| 5.1 | Diagram of Procedures | |
| 5.2 | Subject Preparation | |
| 5.3 | Description of Study Procedures | |
| 5.4 | Follow-up | |
| | udy Data Collection and Assessments | |
| 6.1 | Image Acquisition Data | |
| 6.2 | Image Attribute Review Data | |
| 6.3 | Safety Assessments | |
| 7. Ou | ıalification and Training Plan | |
| 7.1 | Staff Qualifications | |
| 7.2 | Training Plan for the Protocol and Research Product | |
| | fety | |
| 8.1 | Anticipated Adverse Events | |
| 8.2 | Adverse Event Definitions | |
| 8.3 | Documentation of Safety Events | |
| 8.4 | Reporting of Safety Events and Device Deficiencies/Complaints | |
| 8.5 | Device Deficiencies/Complaints | |
| 9. Eth | nical Conduct of the Study | |
| 9.1 | Ethics Committee | 26 |
| 9.2 | Regulatory Agencies and Competent Authority(ies) | |
| 9.3 | Management of Protocol Modifications and Amendments | 26 |

**Study Title:** Patient-Assisted Compression – Impact on Image Quality and Workflow **Study No:** 124.03-2017-GES-0002



| 9.4 | Participant Information and Informed Consent | 26 |
|---|---|---|
| 9.5 | Early Termination of the Study | |
| 10. Sta | tistical Methods | |
| 10.1 | Statistical Hypothesis | 27 |
| 10.2 | Sample Size Determination | |
| 10.3 | Statistical Analysis | |
| 10.4 | Handling of Missing Data | |
| 10.5 | Deviation(s) from the Original Statistical Methods | |
| 11. Qu | ality Assurance and Control | |
| 11.1 | Data Management | |
| 12. Moi | nitoring Plan | |
| 12.1 | Confidentiality and Data Protection | |
| 12.2 | Publication Pólicy | |
| Referer | nces | |
| | dix A – STUDY SCHEDULE | |
| | dix B – Study Site and Investigator List | |
| List o | f Figures and Tables | |
| • | . –Senographe Pristina mammography device with remote control for patien | · |
| Figure 2 | ${f 2}$ – Schematic showing image acquisitions based on the randomly-assigned ${f 1}$ | preast of interest (i.e. first o |
| second l | breast) | 18 |
| Figure 3 | 5 – Diagram of study procedures. | 19 |
| • | 1 - Schedule of Study Procedures | 37 |

**Study No:** 124.03-2017-GES-0002



### **DOCUMENT AND VERSION CONTROL**

This section records all changes made to the protocol for a specific study. In the table below, record every relevant change by indicating what changes were made.

| Revision | Date | Revision Author | Comments/Changes |
|---|---|---|---|
| 1.0 | 22/May/2017 | Carrie Lauer | Clinical Writer – This is the initial version. |

**Study No:** 124.03-2017-GES-0002



#### LIST OF ABBREVIATIONS AND TERMS

2D Two dimensional
 3D Three dimensional
 AE Adverse Event
 ADE Adverse Device Effect

ALARP As Low as Reasonably Practicable

CA Competent Authority

CAPM GE Clinical Affairs Project Manager

CC Craniocaudal

CCG Case Report Form Completion Guidelines

CFR Code of Federal Regulations

CHF Clinical History File (synonymous with e-Trial Master File)

CRF Case Report Form

DBT Digital Breast Tomosynthesis
DCF Data Clarification Form
EC Ethics Committee
EU European Union

FDA United States Food and Drug Administration

FFDM Full-field Digital Mammography

GCP Good Clinical Practice (see ISO 14155:2011) <sup>1</sup>

GE General Electric

GEHC General Electric Healthcare

Guidance Guidance for Industry and FDA Staff - Class II Special Controls Guidance Document: Full-Field Digital

Mammography System (2012)

ICF Informed Consent Form

ISO International Standards Organization

MLO Mediolateral Oblique

MQSA Mammography Quality Standards Act

MWS GE MyWorkshop Internal Documentation System

PA Patient-assisted PI Principal Investigator

Reader Interpreting Physician, as defined under U.S. FDA 21CFR §900.12(a)(1)(i)(B)(2)

SADE Serious Adverse Device Effect

SAE Serious Adverse Event TC Technologist-controlled

US United States

USADE Unexpected Serious Adverse Device Effect

**Study Title:** Patient-Assisted Compression – Impact on Image Quality and Workflow **Study No:** 124.03-2017-GES-0002



| STUDY SYNOPSIS | |
|---|---|
| Sponsor: | General Electric Company, acting through its GE Healthcare Business |
| Research Type: | This is a Clinical, single-blind, randomized, prospective research study. |
| Regulatory Status: | This is a pre-market research study of the following products: Pre-market: Patient-assisted compression on Senographe Pristina Post-market: Technologist-controlled compression on Senographe Pristina |
| Background and<br>Rationale: | Patient-assisted compression allows the patient to participate in controlling the amount of compression force during mammography and is a personalized approach that has demonstrated successful reduction in discomfort experienced during mammography. GE Healthcare's Senographe Pristina, an innovative mammography platform that provides both two-dimensional (2D) and three-dimensional (3D) imaging capabilities, offers both standard and patient-assisted compression modes. This study is being conducted to compare the image quality of breast images obtained using standard compression and patient-assisted (PA) compression, and to evaluate the impact of patient-assisted compression on clinical workflow. Results from this study are intended to support regulatory submissions. |

**Study No:** 124.03-2017-GES-0002



#### Procedures/ Methods:

The study population will consist of adult asymptomatic women presenting for screening 2D mammography. One breast of each subject will be identified as the "breast of interest," which will undergo two-view (craniocaudal and mediolateral oblique) PA compression and image acquisition, immediately followed by technologist-controlled (TC) compression and image acquisition. The breast of interest will be randomly assigned to either the first breast imaged during the exam or the second breast imaged. TC compression and imaging, and procedures performed on the subject's other breast will be conducted per standard of care.

Following image acquisition, image quality evaluation will be conducted by MQSA-qualified readers. Prior to the reading session, images will be de-identified and the following information will be removed from the DICOM header to blind readers to the compression mode used during acquisition: time stamp, compression force, and breast thickness. Two (2) readers will evaluate each PA and TC compression image set collected from each subject's breast of interest and assess the acceptability of image attributes, as defined in the *Guidance for Industry and FDA Staff - Class II Special Controls Guidance Document: Full-Field Digital Mammography System* (2012). A third reader will provide adjudication, if there is disagreement for a given image set's overall clinical image quality.

Workflow data, including time to complete image acquisition for each compression mode and the incidence of technologist intervention during acquisition, will also be collected.

The proportion of PA image sets that are of equal or higher acceptability than TC image sets will be calculated. A 95% confidence interval will be calculated using asymptotic method with continuity correction. The proportion of image sets indicated for repeated image acquisition when using PA mode or TC mode will be summarized. Other endpoint data will be summarized using descriptive statistics. No statistical hypothesis is being tested in this study.

#### Objectives:

The **primary objective** is to compare the acceptability of overall image quality in unilateral two-view (CC and MLO) breast images acquired using PA and TC compression modes.

#### The **secondary objectives** are:

- To evaluate the need for repeat image acquisition when using PA and TC compression modes: and
- To evaluate acceptability of mammographic attributes for unilateral twoview breast images acquired using PA and TC compression modes, per the Guidance for Industry and FDA Staff - Class II Special Controls Guidance Document: Full-Field Digital Mammography System (2012; hereafter referred to as the "Guidance").

#### The **exploratory objectives** are:

- To collect workflow data for PA compression and TC compression, and
- To collect breast thickness, radiation dose, and compression force for images acquired using PA and TC compression.

**Study No:** 124.03-2017-GES-0002



#### **Endpoints:**

The **primary endpoint** is the overall image quality acceptability on a per subjectbasis using a binary response of either acceptable or unacceptable for unilateral, two-view PA and TC compression image sets.

#### The secondary endpoints are:

- Number of incidences per image set when the technologist and/or readers indicate a repeat acquisition for PA and TC compression; and
- Acceptability of mammographic attributes, as defined in the *Guidance* and as described in Section 6.2 Image Attribute Review Data.

The **exploratory endpoints** will be collected per subject for each study-specific PA and TC compression. The endpoints are:

- Time to complete image acquisition;
- Type and incidence of technologist interventions (e.g. technologist uses footswitch to increase compression); and
- Breast thickness, radiation dose, and compression force.

The **safety endpoints** are the type and number of AEs, SAEs, and device issues

#### Eligibility criteria:

#### Inclusion criteria:

- 1) Are women aged 40 years or older;
- Are asymptomatic and scheduled for FFDM screening mammography;
- 3) Have left and right breasts;
- 4) Have breast sizes compatible with the dimensions of a 24 x 31 cm image detector, without anatomical cut-off;
- Are documented as non-pregnant based on the investigator's medical judgment and in consideration of local clinical practice standards for evidence of non-pregnancy;
- 6) Are able and willing to comply with study procedures; and
- 7) Are able and willing to provide written informed consent to participate.

#### Exclusion criteria:

- Have been previously included in this study or are participating in another study expected to interfere with study procedures or outcomes;
- 2) Have undergone diagnostic or surgical intervention(s) or procedure(s) on either breast, including breast biopsy, lumpectomy, or reconstruction, within five (5) years (≤ 5 years) of the study exam date;
- 3) Are currently undergoing radiotherapy or chemotherapy, or have a history of prior radiotherapy treatment on either breast;
- 4) Are currently lactating; or
- 5) Have breast implants.

**Study Title:** Patient-Assisted Compression – Impact on Image Quality and Workflow **Study No:** 124.03-2017-GES-0002



| Sample size and Sites: | Up to 36 subjects from one (1) site will be included as part of this study to achieve the targeted number of complete and evaluable subjects. The target sample size for this study is 30 subjects, providing 60 evaluable image sets for the image attribute review (30 PA compression image sets and 30 TC compression image sets). The number of subjects was determined based on Sponsor discussions with a U.S. FDA Medical Officer, who indicated that, during MQSA re-accreditation, sites are requested to submit sample images. If an issue is identified with the sample images, an Advanced Mammographic Review occurs, where the quality of 30 images is assessed to determine whether the issue was isolated or systemic. |
|---|---|
| Study duration: | The study is expected to last approximately three (3) months. |

**Study Title:** Patient-Assisted Compression – Impact on Image Quality and Workflow **Study No:** 124.03-2017-GES-0002



| ADMINISTRATIVE STRUCTURE OF INVESTIGATION | | |
|---|---|---|
| Clinical Affairs | Sara Lam | GE Healthcare (GEHC) |
| Project Manager | Tel: 1-262-548-2369 | Address: 3000 N Grandview Blvd |
| (Sponsor Contact): | e-mail: Sara.J.Lam@ge.com | Waukesha, WI 53188 U.S. |
| Research Manager: | Sandhya Parameswaran | GEHC |
| | Tel: 1-262-951-8169 | Address: 3000 N Grandview Blvd |
| | e-mail: Sandhya.Parameswaran@med.ge.com | Waukesha, WI 53188 U.S. |
| Medical Monitor: | Ron von Jako, MD, PhD | GEHC |
| ricarcari formor. | Tel: 1-617-669-3200 | Address: 1100 Technology Park Drive |
| | e-mail: Ron.VonJako@med.ge.com | Billerica, MA 01821 U.S. |
| Biostatistician: | Keyi Wang | GEHC |
| | Tel: 1-262-548-2945 | Address: 3000 N Grandview Blvd |
| | <i>e-mail</i> : Keyi.Wang@ge.com | Waukesha, WI 53188 U.S. |

**Study No:** 124.03-2017-GES-0002



### 1. BACKGROUND AND JUSTIFICATION

### 1.1 Screening Mammography and Patient-Assisted Compression

Leading authorities on breast cancer recommend regular screening mammography for women aged 40 years and older as a means of early detection for breast cancer, leading to increased survival rates and more treatment options. <sup>2, 3, 4</sup> Numerous randomized trials have demonstrated that regular mammographic screening reduces breast cancer mortality, <sup>5, 6, 7, 8, 9</sup> with more than 40% reduction in breast cancer deaths. <sup>10, 11</sup> Amidst the success of screening mammography, clinicians struggle to maintain patient participation in regular screening programs. Notably, a systematic review by Whelehan, et al. concluded that pain experienced during screening mammography (e.g. compression pain) contributed to reduced rates of repeat participation in regular screening programs. <sup>12</sup>

Adequate breast compression during mammography creates uniform thickness and flattens tissues, <sup>4</sup> which is necessary to obtain sufficient image quality <sup>4, 13, 14</sup> and reduce radiation dose. <sup>4, 15</sup> Various methods are being investigated to maintain sufficient compression while reducing pain associated with mammography. Specifically, studies have shown that a personalized approach to compression can significantly reduce pain intensity and discomfort experienced by patients while maintaining diagnostic image quality. <sup>16, 17, 18</sup>

Patient-controlled compression allows the patient to control the amount of compression force during mammography and is a personalized approach that has demonstrated successful pain reduction in mammography. <sup>16</sup> GE Healthcare's Senographe Pristina, an innovative mammography platform that provides both two-dimensional (2D) and three-dimensional (3D) imaging capabilities, offers standard and patient-assisted compression modes. The study described herein is being conducted to compare the image quality of breast images obtained using standard compression and patient-assisted compression in an asymptomatic female population undergoing full-field digital (FFDM) 2D screening mammography. This study will also evaluate the impact of patient-assisted compression on clinical workflow. Results from this study are intended to support regulatory submissions.

#### 1.2 Controls and Minimization of Bias

Due to the inherent difference in utility of standard and patient-assisted compression modes, study subjects and study staff will not be blinded to the compression mode. However, the following bias control methods will be employed in this study:

- Selection bias will be limited by consecutively enrolling eligible subjects.
- Spectrum bias will be limited by using a population expected to represent the general population at the investigational site, without regard to race or ethnicity.
- Patient-assisted compression will be randomly assigned to either the first or second breast imaged to mitigate subject-learning bias associated with the amount of compression required for image acquisition.
- Readers conducting image quality evaluations will be blinded to the compression mode used to obtain the images.
- A minimum of three (3) radiology technologists will conduct the study procedures to mitigate bias introduced by technologist-specific practices.



### 2. DEVICE/PRODUCT DESCRIPTION

# 2.1 Identity, Mechanism, and Function of Investigational Device

Name: Patient-Assisted Compression, Senographe Pristina

Modality/Type: Imaging, Women's Health

Manufacturer: GE

**Software version**: Senographe Pristina 1.0, Axis version 1.50

**Regulatory Status**: Pre-market

**Note**: A record of number of products issued, along with applicable identification numbers (e.g. serial/lot/batch) and components/accessories used in this study will be retained by the Sponsor as part of the clinical history file (CHF), as required by applicable laws and regulations.

Patient-Assisted Compression, Senographe Pristina (Figure 1) is a commercial mammography medical device consisting of the Senographe Pristina FFDM system (2D) and Senographe Pristina DBT option (3D). The platform is an evolution of the cleared/approved Senographe Essential FFDM system (2D) and SenoClaire DBT option (3D). Senographe Pristina includes the same clinical applications as traditional mammography systems and is designed to improve workflow while maintaining imaging capabilities and image quality of FFDM and DBT breast imaging. The FFDM option will be used for the purposes of this study.

Senographe Pristina includes the hardware and software components required for multi-modality functioning and is designed to improve patient experience, patient throughput, and radiographer experience. The system offers two compression modes – standard mode and the optional patient-assisted compression mode (referred to as "PA compression" hereafter). The patient-assisted feature enables the patient to personally refine breast compression using a hand-held remote control (Figure 1) after the compression has been initiated by the operator, which is required to ensure proper breast positioning.



Figure 1 – Senographe Pristina mammography device with remote control for patient-assisted compression mode.

The research device (i.e. Senographe Pristina with PA compression), instructions for use, or packaging shall indicate that the research device is for use in a research investigation, in accordance with applicable regulations in the U.S., including U.S. FDA 21 CFR and other applicable laws and regulations. Senographe Pristina with PA compression will be exclusively used for research purposes.



The results of this study are intended to support regulatory submissions for PA compression. Results may be used to help commercialize the product in other global regions in the future, at the discretion of the Sponsor.

### 2.2 Mammography Review Workstation

An FDA-cleared mammography review workstation or other image review system will be used in this study to display images during reader evaluations of the image sets. Review workstations/systems are not a component of Senographe Pristina.

The study-specific images will be labelled for research use only, and the investigational image sets will be exclusively used for research purposes.

#### 2.3 Intended Use

Senographe Pristina is intended to be used for screening and diagnostic mammography; however, screening mammography is the focus of this study. Study procedures are intended for research purposes and are not intended as a substitute for required medical care.

### 2.4 Comparator

The comparator is the technologist-controlled compression mode of Senographe Pristina (referred to as "TC compression" hereafter). This is considered the "standard" compression mode, which is currently cleared for use with Senographe Pristina.

# 2.5 Concomitant/Ancillary Administrations

### 2.5.1 Medications and Biologic Products

No medications or biologic products will be administered as part of study procedures.

#### 2.5.2 Laboratory Tests and Sample Processing

No laboratory tests or sample processing is planned as part of the study procedures.

# 2.6 Accountability

Accurate and adequate records will be maintained for all devices/products, from time of shipment to the site until return or disposal of all devices issued by the Sponsor as part of this study, as required by applicable laws and regulations. The Principal Investigator (PI) will be ultimately responsible for the security and integrity of research devices/products at the investigational site during the study.

#### 2.6.1 Issuance

The PA compression product will be provided by the Sponsor while the Senographe Pristina and the review workstations will be provided by the site. Calibration/maintenance of study product(s) is not planned to maintain integrity of study data.

#### 2.6.2 Disposition

Product(s) provided to the site by the Sponsor will be returned to the Sponsor, in accordance with applicable laws and regulations.

 GE MWS DOC1991348 Ver: 1.0; 22/May/2017

**Study No:** 124.03-2017-GES-0002



# 2.7 Anticipated Risks and Benefits

The device under study has undergone risk assessment, in accordance with International Standards Organization (ISO) 14971:2012. Risks have been mitigated to levels as low as reasonably possible (ALARP) and are not expected to exceed risks associated with the routine clinical breast cancer screening procedures that the subject has been prescribed outside of the study. The operator's manual highlights warnings, cautions, and potential conventional risks associated with the exam.

Breast imaging procedures will be conducted using post-market Senographe Pristina systems with pre-market PA compression mode installed. Breast imaging procedures will be conducted per the site's standard of care, with the exception of the investigational imaging, which will consist of unilateral two-view (craniocaudal [CC] and mediolateral oblique [MLO]) imaging acquired using the PA compression. There will be no repeat imaging administered using PA compression mode.

No additional medications will be administered beyond those regularly required for the subject's medical care outside of this study, and regular medication should not be adversely impacted or delayed by study participation. Post-trial care and follow-up are not required by this study.

There is no expected benefit to study subjects participating in this research. The results of this study may benefit future patients by increasing knowledge about the PA compression mode of Senographe Pristina.

### 2.7.1 Risk Category and Rationale

The Senographe Pristina FFDM system with PA compression mode, as used in this study, is not considered a significant risk device per the 21 CFR §812.3 definition:

- 1) it is not intended as an implant;
- 2) is not purported or represented to be for a use in supporting or sustaining human life;
- 3) is not for a use of substantial importance in diagnosing, curing, mitigating, or treating disease, or otherwise preventing impairment of human health; and
- 4) it does not otherwise present a potential for serious risk to the health, safety, or welfare of a subject.

This designation of non-significant risk is supported by the study design, in which the data obtained will not be used as the sole measure of diagnosis without distinct confirmation from conventional methods, such as mammography on an approved/cleared device or other standard of care procedures at the investigational site.

#### 3. STUDY OBJECTIVES AND ENDPOINTS

# 3.1 Purpose of the Study

The purpose of this study is to collect clinical evidence associated with image quality and workflow to support regulatory submissions for Senographe Pristina PA compression mode.

### 3.1.1 Primary Objective

The primary objective is to compare the acceptability of overall image quality in unilateral two-view (CC and MLO) breast images acquired using PA and TC compression modes.

### 3.1.2 Secondary Objectives

The secondary objectives are:

- To evaluate the need for repeat image acquisition when using PA and TC compression modes; and
- To evaluate acceptability of mammographic attributes for unilateral two-view breast images acquired using PA and TC compression modes, per the Guidance for Industry and FDA Staff - Class II Special

 GE MWS DOC1991348 Ver: 1.0; 22/May/2017



Controls Guidance Document: Full-Field Digital Mammography System (2012; hereafter referred to as the "Guidance").

### 3.1.3 Exploratory Objectives

The exploratory objectives are:

- To collect workflow data for PA compression and TC compression, and
- To collect breast thickness, radiation dose, and compression force for images acquired using PA and TC compression.

### 3.1.4 Safety Objective

The objective is to collect safety information, including adverse events (AEs), serious adverse events (SAEs), and product issues.

### 3.2 Study Endpoints

### 3.2.1 Primary Endpoint

The primary endpoint is the overall image quality acceptability on a per subject-basis using a binary response of either acceptable or unacceptable for unilateral, two-view PA and TC compression image sets.

### 3.2.2 Secondary Endpoints

The secondary endpoints are:

- Number of incidences per image set when the technologist and/or readers indicate a repeat acquisition for PA and TC compression; and
- Acceptability of mammographic attributes, as defined in the *Guidance* and as described in Section 6.2 Image Attribute Review Data.

#### 3.2.3 Exploratory Endpoints

The exploratory endpoints will be collected per subject for each study-specific PA and TC compression. The endpoints are:

- Time to complete image acquisition;
- Type and incidence of technologist interventions (e.g. technologist uses footswitch to increase compression); and
- Breast thickness, radiation dose, and compression force.

#### 3.2.4 Safety Endpoints

The safety endpoints are the type and number of AEs, SAEs, and device issues.

# 3.3 Summary of Study Design

This is a pre-market, Clinical, single-blind, prospective, randomized research study conducted at one (1) site in the U.S.

 GE MWS DOC1991348 Ver: 1.0; 22/May/2017



#### 4. STUDY DESIGN

### 4.1 Study Population

The study population will consist of asymptomatic adult women presenting for screening FFDM breast imaging, which is representative of the general population expected to use Senographe Pristina in clinical practice.

# 4.2 Number Subjects

Up to 36 subjects will be enrolled into this study at one (1) site to achieve the targeted number of 30 complete and evaluable subjects.

# 4.3 Protection of Vulnerable Subjects

Vulnerable subjects are individuals whose willingness to volunteer in a clinical investigation could be unduly influenced by the expectation, whether justified or not, of benefits associated with participation or of retaliatory response from senior members of a hierarchy in case of refusal to participate.

The Sponsor shall avoid improper influence on, or inducement of, the subject, monitor, any investigator(s), or other parties participating in, or contributing to, the clinical investigation.

All investigators shall avoid improper influence on, or inducement of, the subject, Sponsor, monitor, other investigator(s), or other parties participating in, or contributing to, the clinical investigation.

This study does not examine any groups of subjects who are considered to be vulnerable subjects in the country in which the study is being conducted.

# 4.4 Eligibility Criteria

#### 4.4.1 Inclusion Criteria

Subjects who meet all the following inclusion criteria may be included:

- 1) Are women aged 40 years or older;
- 2) Are asymptomatic and scheduled for FFDM screening mammography;
- 3) Have left and right breasts;
- 4) Have breast sizes compatible with the dimensions of a  $24 \times 31$  cm image detector, without anatomical cut-off;
- 5) Are documented as non-pregnant based on the investigator's medical judgment and in consideration of local clinical practice standards for evidence of non-pregnancy;
- 6) Are able and willing to comply with study procedures; and
- 7) Are able and willing to provide written informed consent to participate.

#### 4.4.2 Exclusion Criteria

- 1) Have been previously included in this study or are participating in another study expected to interfere with study procedures or outcomes;
- 2) Have undergone diagnostic or surgical intervention(s) or procedure(s) on either breast, including breast biopsy, lumpectomy, or reconstruction, within five (5) years (≤ 5 years) of the study exam date;

**Study No:** 124.03-2017-GES-0002



- Are currently undergoing radiotherapy or chemotherapy, or have a history of prior radiotherapy treatment on either breast;
- 4) Are currently lactating; or
- 5) Have breast implants.

# 4.5 Recruiting and Screening

Subjects will be recruited for potential enrollment into this study from an adult asymptomatic female population scheduled for screening FFDM at the site. Subjects will be screened for enrollment against the inclusion and exclusion criteria, and enrollment determinations will be made by the PI. Recruitment, screening, and enrollment will be conducted per the standard procedures of the investigational site. All subject participation will be voluntary.

Following recruitment, a subject will be considered enrolled (the point of enrollment) once she signs and dates the informed consent form (ICF). Once enrolled, the subject will be assigned a unique subject number, which will not contain information that could identify her (e.g. subject name or date of birth). The unique subject number will be used to label case report form (CRF) data for the subject throughout her participation in the study.

#### 4.6 Breast of Interest Randomization

One (1) breast per subject will undergo study-specific procedures (hereafter referred to as "breast of interest") while the second breast will be imaged per standard of care. The breast of interest will be randomized across all subjects so that approximately half the subjects will be assigned to the first imaged breast and the other half will be assigned to the second imaged breast (Figure 2).

Site technologists conducting the study will perform each subject's mammography exam per standard practice. Thus, the laterality of the breast of interest will solely depend on which breast (left or right) the technologist images first and second in standard practice.



Figure 2 – Schematic showing image acquisitions based on the randomly-assigned breast of interest (i.e. first or second breast).

#### 4.7 Criteria for Withdrawal/Discontinuation

A subject may withdraw from study participation at any time, for any reason, and the investigator may withdraw a subject at any time, for any reason. The reasons for withdrawal and discontinuation for any subject shall be recorded on a case report form (CRF) and reported to the Sponsor. The Ethics Committee (EC) should be notified per their notification-of-subject-withdrawal policy.

 GE MWS DOC1991348 Ver: 1.0; 22/May/2017



A subject shall be withdrawn from the study if a study-related PA compression in either CC or MLO view is not completed (i.e. no image is acquired due to inadequate compression or positioning). If a subject withdraws or is withdrawn, all efforts will be made to complete and report study data up to the time of withdrawal. A complete final evaluation at the time of the subject's withdrawal shall be made and recorded on a CRF. If the reason for withdrawal is related to an adverse event (AE) or serious adverse event (SAE), monitoring of the subject will continue until the outcome is evident.

Any data collected for the subject, up until the time of withdrawal or discontinuation, may still be included in the study results and provided to the Sponsor, unless the subject requests that their data not be used. The site shall document all requests by subjects regarding their data use.

### 5. STUDY PROCEDURES

### 5.1 Diagram of Procedures

Figure 3 shows a high-level sequence of study procedures that will be conducted in this study.



Figure 3 - Diagram of study procedures.



# **5.2 Subject Preparation**

Study staff will confirm that the subject is eligible and willing to comply with applicable site requirements prior to starting study procedures. Demographic information, clinical history data, and pregnancy/menopausal status will be collected prior to the mammography exam.

No preparation for the breast imaging exam beyond that usually required by the investigational site is needed before procedures. After consenting, however, the study staff will show the subjects how to use the PA compression mode prior to starting the exam.

# 5.3 Description of Study Procedures

### 5.3.1 Image acquisitions

Each subject will undergo her regularly scheduled FFDM imaging exam per standard practices at the investigational site, with the exception of the study-specific image acquisitions using PA compression. For the breast of interest, PA compression and image acquisition will be conducted first and consist of both CC and MLO views. There shall be no repeat imaging administered using PA compression mode. Following two-view PA compression image acquisition, TC compression and standard of care imaging will be conducted on the same breast/breast of interest. Standard of care will be used for imaging of the subject's other breast.

A minimum of three (3) site technologists will perform the image acquisitions and related study procedures. Study procedures shall not impact the order in which the left and right breasts are imaged during the subjects' exams.

There will be two (2) study-specific <u>image sets</u> of the breast of interest for each subject. Image sets will consist of CC and MLO views obtained using PA compression and CC and MLO views obtained using TC compression.

### 5.3.1.1 Image set acquisition time

Study staff will capture the following times associated with the study procedures:

- 1) Amount of time it took to educate the subject on the PA compression mode and remote control.
- 2) Start time of first PA compression on breast of interest.
- 3) Start time of first TC compression on breast of interest.

#### 5.3.2 Image attribute review

Following acquisition, study-specific images will be de-identified, and the time stamp, compression force, and breast thickness will be removed from the DICOM header to ensure the readers are blinded to the compression mode used for each image set.

PA and TC compression image sets will be evaluated by two (2) MQSA-qualified readers, with a third reader to provide adjudication if disagreement is observed between the two (2) readers' evaluations of "overall clinical image quality" (i.e. item number 9 in Section 5.3.2 Image attribute review). Images will be displayed on site-provided mammography review workstations/systems in the order in which they were acquired from the study subjects. Each reader will evaluate each image set independently from other reader(s) and have the freedom to navigate between views, as he/she would do in clinical practice.

In addition to the images, the following case data will be available to the readers for each image set during image attribute review:

- Techniques (anode, filter, kVp, mAs, half-value layer)
- Estimated average glandular dose per view (mGy)



# 5.4 Follow-up

No follow-up will be conducted in this study.

#### 6. STUDY DATA COLLECTION AND ASSESSMENTS

### 6.1 Image Acquisition Data

The following data will be collected on a study CRF during the mammography exams:

- 1) Date of mammography exam
- 2) Demographic information, including age and ethnicity
- 3) Menopausal status
- 4) Size of paddle used for imaging (per breast)  $24 \times 29.8$  cm or  $19 \times 23$  cm
- 5) Time to educate patient of PA compression 1-2 minutes, 3-5 minutes, or more than 5 minutes
- 6) Breast of interest First breast imaged or Second breast imaged
- 7) Laterality of the breast of interest Right or Left
- 8) Start time of first PA compression on breast of interest (hh:mm) <sup>1</sup>
- 9) Start time of first TC compression on breast of interest (hh:mm) 1

When a subject's mammography exam is complete, the following data will be collected on a study CRF:

- 1) Considering the PA compression only, did the technologist intervene while the subject was controlling the compression? Yes or No. If yes, please indicate which of the following interventions were done:
  - a. Use footswitch to increase compression
  - b. Used footswitch to decrease compression
  - c. Used manual knobs to increase compression
  - d. Used manual knobs to decrease compression
- 2) Considering the <u>PA compression only</u>, would you have repeated the image acquisition? Yes or No. If yes, please select the option below that best describes the reasoning.
  - a. Positioning
  - b. Compression
  - c. Other, please explain.
- 3) Considering the <u>TC compression only</u>, did you repeat image acquisition? Yes or No. If yes, please select the option below that best describes the reasoning.
  - a. Positioning
  - b. Compression
  - c. Other, please explain.
- 4) Compression force (daN) obtained from DICOM header
- 5) Breast thickness (mm) obtained from DICOM header

GE MWS DOC1991348 Ver: 1.0; 22/May/2017

GE Healthcare - Confidential

<sup>&</sup>lt;sup>1</sup> End times will be retrieved from the DICOM header of the last image acquired for a given image set.



- 6) AGD (mGy) obtained from DICOM header
- 7) Per-view acquisition parameters (mAs and kVp) obtained from DICOM header

# 6.2 Image Attribute Review Data

Following training (see Section 7. Qualification and Training Plan), readers will evaluate all image sets from all cases by classifying each of the following image attributes as either "Acceptable" or "Not Acceptable" on CRFs.

- 1) Breast positioning, assessing coverage of the breast on craniocaudal and mediolateral oblique view, separately
- 2) Exposure, assessing visualization of the adipose and fibroglandular tissues, and visualization of breast tissue underlying the pectoralis muscle, separately
- 3) Breast compression, assessing overlapping breast structures, uniformity of exposure of fibroglandular tissues, adequacy of penetration of thicker portions of the breast, exposure of thinner areas, and motion unsharpness
- 4) Image contrast for differentiation of subtle tissue density differences
- 5) Sharpness, assessing the edges of fine linear structures, tissue borders, and benign calcifications
- 6) Tissue visibility at the skin line
- 7) Noise, i.e., noise obscuring breast structures or suggestive of structures not actually present
- 8) Artifacts due to image processing, detector failure and other factors external to the breast on hard-copy and soft-copy displays
- 9) Overall clinical image quality
  - a. If you answered "not acceptable" for overall clinical image quality, would you request repeat imaging in standard clinical practice? Yes or No.
  - b. If yes, which view would you request for repeat imaging? CC only, MLO only, or both CC and MLO?

If an issue is encountered by any reader during the image attribute review of any image set, an explanation of the issue will be documented on a CRF by the reader.

Readers will also classify the breast density of each image set as follows:

- 1) Almost entirely fatty
- 2) Scattered areas of fibroglandular density
- 3) Heterogeneously dense
- 4) Extremely dense

# 6.3 Safety Assessments

The description, severity, and device relatedness of any AE or SAE during the study will be recorded. Subjects will, if necessary, be provided with emergency care. In the event of any device issues, the event will be recorded. Safety reporting will be conducted as described in this protocol.



### 7. QUALIFICATION AND TRAINING PLAN

# 7.1 Staff Qualifications

All members of the study staff participating in the conduct of the clinical investigation shall be qualified by education, training and/or experience to perform their tasks, and this shall be documented appropriately, as per ISO 14155:2011. Specifically, readers shall be MQSA-qualified.

# 7.2 Training Plan for the Protocol and Research Product

Before starting the study, study staff will be trained on the requirements and procedures set forth in this study protocol, including completion of ICFs, CRFs, and other study documentation. Training will also be provided to ensure appropriate storage and handling of data, and all study staff will be required to be trained on Good Clinical Practice (GCP) guidelines per ISO 14155: 2011.

A record of all formal training will be stored in the Site Regulatory Binder and provided to the Sponsor for inclusion in the Sponsor's CHF. Documentation of training will include:

- Title of Training
- Training objectives
- Training logistics (trainer and training methods)
- Documentation of trainees
- Training content (e.g. device operation, protocol review and CRF completion)

Study staff directly operating the PA compression product will be qualified based on mammographic experience and trained to use PA compression by a GE application specialist.

The Principal Investigator will be ultimately responsible for execution of this study in accordance with the protocol and for device use in this study by members of the study staff.

#### 8. SAFETY

# 8.1 Anticipated Adverse Events

Mammography is an x-ray examination of the breasts. As with all x-ray exams, mammography involves ionizing radiation. The amount of radiation from a standard FFDM mammography exam, even with the addition of the study-specific unilateral, two-view imaging, is small and equal in cancer risk to the total body radiation received naturally from the environment over a period of a few months.

There are no known additional medical risks or side effects from Senographe Pristina FFDM with PA compression mode beyond those of similar conventional clinical procedures on other commercial mammography devices. Foreseeable AEs that apply to mammography and are also applicable to digital mammography using the Senographe Pristina with PA compression mode may include, but are not limited to:

- Bruising (uncommon);
- Skin irritation (uncommon), abrasions (uncommon), or tears (rare);
- Discomfort (common).

The study staff conducting the research is trained to recognize these reactions, and should it be necessary, other medical care is available at the site. Subjects will be followed for AEs from the time they enter the imaging suite for their exam until the time they exit the imaging suite after the exam.

**Study No:** 124.03-2017-GES-0002



It is generally agreed that the risk to a fetus from radiation in a screening mammography exam is minimal <sup>19</sup>; however, it is standard clinical practice to try to determine pregnancy status of women referred for mammography and not allow women known or suspected to be pregnant to undergo screening mammography or other elective radiologic procedures.

There is always a chance of unexpected risks. Throughout the study, the Sponsor will evaluate and update safety information in study documents.

### 8.2 Adverse Event Definitions

**Adverse Event (AE)**: any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device [ISO 14155:2011 3.2]. This includes events related to the investigational device or the comparator and to the procedures involved. For users or other persons, this is restricted to events related to the investigational medical device.

**Serious Adverse Event (SAE)**: an adverse event that led to death; led to a serious deterioration in the health of the subject, that either resulted in a life-threatening illness or injury, a permanent impairment of a body structure or a body function, or in-patient or prolonged hospitalization, or medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to body structure or a body function; or led to fetal distress, fetal death or a congenital abnormality or birth defect. Planned hospitalization for a pre-existing condition, or a procedure required by the protocol without serious deterioration in health, is not considered a SAE [ISO 14155:2011 3.37].

**Adverse Device Effect (ADE)**: an adverse event related to the use of an investigational medical device [ISO 14155:2011 3.1]. This includes any adverse events resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the investigational medical device. This includes any event that is a result of a user error or intentional misuse of the investigational device [ISO 14155:2011 3.43].

**Serious Adverse Device Effect (SADE)**: an adverse device effect that has resulted in any of the consequences characteristic of a serious adverse event [ISO 14155:2011 3.36].

**Device deficiency:** an inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety, or performance, such as malfunctions, use errors, and inadequate labelling [ISO 14155:2011 3.15].

**Unanticipated serious adverse device effect (USADE):** a serious adverse device effect, which by its nature, incidence, severity, or outcome has not been identified in the current version of the risk analysis report [ISO 14155:2011 3.42]. In the United States, any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, a device, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the study documents, will be reported in accordance with 21 CFR §812.3 and applicable laws and regulations.

# 8.3 Documentation of Safety Events

All adverse events (AE), including all serious adverse events (SAE), are required to be collected, investigated, and documented during the study reporting period, as defined in the study procedure set forth in this protocol. Documentation will include:

- Description of Event
- Date of onset and resolution
- Severity (mild, moderate, or severe)
  - Mild: Symptom(s) barely noticeable to the subject or does not make the subject uncomfortable.
     The AE does not influence performance or functioning. Prescription drugs are not ordinarily needed for relief of symptom(s).

 GE MWS DOC1991348 Ver: 1.0; 22/May/2017 Study No: 124.03-2017-GES-0002



- Moderate: Symptom(s) of a sufficient severity to make the subject uncomfortable. Performance
  of daily activities is influenced. Treatment of symptom(s) may be needed.
- Severe: Symptom(s) of a sufficient severity to cause the subject severe discomfort. Treatment for symptom(s) may be given.
- Serious (yes/no)
- Causal relationship to investigational medical device? (not related, possibly related, or related)
  - Not related: The adverse event is reasonably expected to be related to (or caused by) a
    concurrent illness, effect of another device/drug or other cause, and is unlikely related to the
    investigational product.
  - Possibly related: The adverse event is reasonably expected to be related to the investigational product, and an alternative etiology is equally or less likely compared to the potential relationship to investigational product.
  - Related: There is a strong relationship to investigational product or recurs on re-challenge, and another etiology is unlikely or there is no other reasonable medical explanation for the event.
- Treatment given and/or action taken (procedure stopped, withdrawn from study, or no action)
- Anticipated (yes/no)

# 8.4 Reporting of Safety Events and Device Deficiencies/Complaints

The following events are to be reported to the Sponsor within 72 hours of the event occurrence and to the EC per their policy:

- All SAEs and USADEs
- All device issues that could possible lead to an SAE

Additional follow-up information may be requested by the Sponsor. In addition, safety information may be shared with regulatory agencies and other participating sites, as required by applicable law and regulation.

If the event resulted in the death of a subject, the event shall also be reported via telephone to the Sponsor within 24 hours of knowledge of the event. SAEs will be reported to the local EC per their policy.

### Sponsor contact for SAEs and UADEs:

Ron von Jako, MD, PhD Fax: 1-800-888-3983 E-mail: SAE@ge.com

# 8.5 Device Deficiencies/Complaints

Device deficiencies/complaints should be reported to the study Sponsor contact identified on the cover page of this protocol. All device deficiencies/complaints will be collected, fully investigated, and documented in the source document and appropriate Sponsor document during the study reporting period. The PI is responsible for notifying the Sponsor in the event that there is any device issue that could potentially lead to a SAE.

#### 9. ETHICAL CONDUCT OF THE STUDY

The study will be carried out in accordance with the protocol and with principles enunciated in the current version of the Declaration of Helsinki; the guidelines of Good Clinical Practice (GCP) for medical devices, as set forth by ISO 14155:2011 and ISO 14971:2012; applicable sections of U.S. FDA 21 Code of Federal Regulations (CFR); and applicable regulatory authority's requirements of the U.S.



The study will be conducted and reported in accordance with applicable policies of the EC and governing regulatory authorities.

#### 9.1 Ethics Committee

The PI will ensure that approval from an appropriately constituted EC is attained for the clinical study prior to enrolling subjects, and Principal Investigator will ensure that documentation of approval is maintained for the duration of the study.

The PI will ensure that the Sponsor is notified of any withdrawal of EC approval within 5 working days of such occurrence. If approval is terminated or suspended, the Principal Investigator will promptly notify the Sponsor and provide written explanation.

# 9.2 Regulatory Agencies and Competent Authority(ies)

The Sponsor will obtain approval from the local regulatory agency and competent authority (CA) before the start of the clinical trial, if necessary, per applicable local laws and regulations. Any additional requirements imposed by the EC or regulatory authority shall be followed, if applicable.

# 9.3 Management of Protocol Modifications and Amendments

Substantial amendments will only be implemented after approval of the EC.

A deviation is any instance(s) of failure to follow, intentionally or unintentionally, the requirements of the protocol. Under emergency circumstances, deviations from the protocol to protect the rights, safety, and wellbeing of human subjects may proceed without prior approval of the Sponsor and the EC/competent authority (CA). Such deviations shall be documented and reported to the Sponsor and the EC as soon as possible. Deviations will be reported as:

- **Critical Deviations:** Deviations that significantly affect the safety, efficacy, integrity, or conduct of the study. These deviations must be reported to the Sponsor no later than 5 working days from awareness of occurrence and reported to the EC per the deviation reporting policy.
- Non-Critical Deviations: Protocol deviations that <u>do not</u> significantly affect the safety, efficacy, integrity, or conduct of the trial. These deviations must be documented on the CRF Protocol Deviation page and will be reviewed by the study monitor.

Non-substantial modifications may be made during the normal course of device optimization, maintenance, and feasibility testing. Non-substantial modifications will be communicated to the CA as soon as possible, if applicable, and to the EC per their policy.

# 9.4 Participant Information and Informed Consent

The investigators will explain to each participant the nature of the study, its purpose, the procedures involved, the expected duration of exposure to the investigational product (if applicable), the potential risks and benefits, and any potential discomforts. Each participant will be informed that participation in the study is voluntary, that she may withdraw from the study at any time, and that withdrawal of consent will not affect her subsequent medical assistance and treatment. The participant must be informed that her medical records may be examined by authorized individuals other than their treating physician.

All participants for the study will be provided an ICF, describing the study and providing sufficient information to allow the participant to make an informed decision about her participation in the study. Informed consent documents will be subject to approval by the EC prior to enrolling subjects in the study.

 GE MWS DOC1991348 Ver: 1.0; 22/May/2017



The participant should read and consider the statement before signing and dating the ICF, and shall be given a copy of the signed document. The ICF must also be signed and dated by the PI (or his/her designee), and it shall be retained as part of the study records.

# 9.5 Early Termination of the Study

The Sponsor may terminate the study prematurely according to certain circumstances. Examples of such circumstances include ethical concerns, insufficient participant recruitment, participant safety concerns, alterations in accepted clinical practice that make the continuation of a clinical trial unwise, early evidence of benefit or harm of the research product, or for any other reason.

#### 10. STATISTICAL METHODS

# 10.1Statistical Hypothesis

No statistical hypothesis is being tested in this study.

# 10.2 Sample Size Determination

The target sample size for this study is 30 subjects, providing 60 evaluable image sets for the image attribute review (30 PA compression image sets and 30 TC compression image sets). The number of subjects was determined based on Sponsor discussions with a U.S. FDA Medical Officer, who indicated that, during MQSA reaccreditation, sites are requested to submit sample images. If an issue is identified with the sample images, an Advanced Mammographic Review occurs, where the quality of 30 images is assessed to determine whether the issue was isolated or systemic.

With a sample size of 30 image pairs, the 95% confidence interval width for the proportion of PA image sets with equal or higher acceptability than TC image sets will be no wider than 13%, when the proportion is 95%.

# 10.3 Statistical Analysis


#### 10.3.1 General Statistical Methods

The study data will be summarized using descriptive statistics. The descriptive statistics for continuous variables will include mean, standard deviation, median, Q1 and Q3, minimum, maximum, and sample size, as appropriate. Categorical variables will be described with counts, percentages, and sample size, as appropriate. A 95% confidence interval may be presented, when necessary.

### 10.3.2 Analysis of Primary Endpoint

The proportion of PA image sets that are of equal or higher acceptability than TC image sets will be calculated. A 95% confidence interval will be calculated using asymptotic method with continuity correction. This analysis will also be performed for subgroups defined by the randomized breast of interest (i.e. breast of interest imaged first versus breast of interest imaged second).

Proportion of images with acceptable overall image quality will be summarized for PA image sets and TC image sets separately, with 95% confidence interval using asymptotic method with continuity correction.

### 10.3.3 Analysis of Secondary and Exploratory Endpoints

The proportion of image sets indicated for repeated image acquisition when using PA mode or TC mode will be summarized. This analysis will also be performed for subgroups defined by the randomized breast of interest.

The acceptability for individual mammographic attributes will be summarized by attribute.

GE MWS DOC1991348 Ver: 1.0; 22/May/2017

**Study No:** 124.03-2017-GES-0002



Time to complete image acquisition for PA mode and TC mode will be summarized descriptively. Type and number of technologist intervention needed during PA mode will be summarized. Similarly, patient characteristics (demographics, breast thickness) and procedural characteristics (radiation dose, compression force) will be summarized using descriptive statistics.

Compression force analysis will also be performed for subgroups defined by the randomized breast of interest.

### 10.3.4 Safety Analysis

AEs, SAEs, and devices issues will be provided in listings and will be summarized descriptively, as deemed necessary.

### 10.3. Interim Analysis

No interim analyses are intended to be conducted as part of this study.

# 10.4 Handling of Missing Data

Analysis will be based on collected data, and no imputation will be done for missing data.

# 10.5 Deviation(s) from the Original Statistical Methods

Any changes or deviations from the original statistical plan specified in this protocol will be described and justified in the final study report per ISO 14155:2011.

### 11. QUALITY ASSURANCE AND CONTROL

# 11.1 Data Management

Data management processes for handling study data will be maintained by the Sponsor.

### 11.1.1 Completion of Case Report Forms (CRFs)

The data reported on the CRFs shall be derived from source documents and be consistent with these source documents. Paper CRFs and/or electronic CRFs (eCRFs) will be used to collect data. The Sponsor will provide e/CRFs and train study staff on completion of e/CRFs using Good Documentation Practices (GDP). CRF Completion Guidelines (CCG) may be provided by the Sponsor to help facilitate training.

e/CRFs are to be completed as information becomes available at the site. e/CRFs should be signed by indicated parties, in indicated area(s), to certify the contents of the form. The Principal Investigator is ultimately responsible for ensuring completion of e/CRFs.

If discrepancies are discovered on paper CRFs during monitoring, the Sponsor's representative will ensure that the study staff makes necessary corrections directly to the CRF(s) prior to collection.

Following CRF collection, the Sponsor will review the data. A Data Clarification Form (DCF) may be provided to the site to correct or clarify discrepancies.

If a site discovers discrepancies after CRF collection, the site may notify the Sponsor and request data modification.

If discrepancies are discovered on the eCRF, whether during monitoring or during data review by the study team, a query will be raised, and the site shall make the correction within the electronic database, noting the reason for change. Data will be considered clean once all queries are answered and closed.

If the Sponsor discovers discrepancies on eCRFs, a query will be raised and necessary corrections will be made by the site. The reason for any changes will be noted. All queries will be resolved prior to study completion.

 GE MWS DOC1991348 Ver: 1.0; 22/May/2017



### 11.1.2 Data Handling and Record Keeping

All documents and data shall be produced and maintained in a manner that assures control and traceability.

#### 11.1.3 Source Data and Documents

Source data includes information in original records, certified copies of original records of clinical findings, observations, or other activities for the study. Source documents for each subject must be retained throughout the investigation, including printed or electronic documents containing source data. Elements should include:

- **Source data and documentation** relevant to data recorded for subject screening and CRF corroboration.
- **Subject records** containing the completed ICFs and CRFs.
- **Regulatory binder** containing the protocol and any subsequent amendments, EC submissions and approvals, blank ICF(s), and site logs.
- **Reference manuals** such as investigator responsibilities, Sponsor, AE/SAE and informed consent guidelines, applicable training materials, and operator manual for PA compression.

The Principal Investigator or institution shall provide direct access to source data during and after the clinical investigation for monitoring, audits, EC review, and regulatory authority inspections.

### 11.1.4 Archiving

All study data must be archived for a minimum of three (3) years after study termination or premature termination of the clinical trial. No source documents or study records will be destroyed without Sponsor notification and approval.

#### 12. MONITORING PLAN

In collaboration with the site, the Sponsor will ensure proper monitoring of the study to confirm that all the research requirements are met. Monitoring visits will oversee the progress of a clinical investigation and ensure that it is conducted, recorded, and reported in accordance with the protocol, written procedures, Good Clinical Practice (GCP) ISO 14155:2011, and the applicable regulatory requirements.

# 12.1 Confidentiality and Data Protection

The investigator affirms and upholds the principle of the participant's right to privacy, and the investigator shall comply with applicable privacy laws. Especially, anonymity of the participants shall be guaranteed when presenting the data at scientific meetings or publishing data in scientific journals.

Individual subject medical information obtained as a result of this study will be considered confidential, and disclosure to third parties will be prohibited. Subject confidentiality will be further ensured by utilizing subject identification code numbers. For data verification purposes, authorized representatives of the Sponsor, a competent authority (CA), or an ethics committee (EC) may require direct access to parts of the medical records relevant to the study, including subject medical history.

### 12.1.1 Storage of Images and Associated Health Data

Images and associated data will be collected and disclosed to the Sponsor as part of this study. Fully de-identified data, which has had all personal identifying information removed, may be stored and used by the Sponsor indefinitely. The Sponsor and/or its authorized representatives may use any de-identified data collected in this study for future technology and engineering development, marketing purposes, education, regulatory submissions, publications, or other possible uses.

 GE MWS DOC1991348 Ver: 1.0; 22/May/2017

**Study No:** 124.03-2017-GES-0002



# 12.2 Publication Policy

The results of this study may be used in future publications. If applicable, the conditions of publication shall be described in a separate contractual agreement.

**Study No:** 124.03-2017-GES-0002



#### REFERENCES

- 1. ISO. Clinical investigation of medical devices for human subjects Good Clinical Practice: International Organization for Standardization; 2011. ISO 14155:2011(E).
- 2. American Cancer Society. *Breast Cancer Facts & Figures 2015-2016*. United States: American Cancer Society; 2015.
- 3. American Cancer Society. Global Cancer Facts & Figures 3rd Edition. Atlanta: American Cancer Society; 2015.
- 4. Nelson HD, Cantor A, Humphrey L, et al. *Screening for Breast Cancer: A Systematic Review to Update the 2009 U.S. Preventive Services Task Force Recommendation*. Rockville: Agency for Healthcare Research and Quality; 2016. 14-05201-EF-1.
- 5. Shapiro S, Strax P, Venet L. Periodic breast cancer screening in reducing mortality from breast cancer. *JAMA*. 1971;215(11):1777-1785.
- 6. Thurfjell E, Lendgren J. Breast cancer survival rates with mammographic screening: similar favorable survival rates for women younger and those older than 50 years. *Radiology*. 1996;201(2).
- 7. Hendrick R, Smith R, Rutledge J, Smart C. Benefit of screening mammography in women aged 40-49: a new meta-analysis of randomized controlled trials. *J Natl Cancer Inst Monogr.* 1997;22:87-92.
- 8. Tabar L, Vitak B, Chen H, Yen M, Duffy S, Smith R. Beyond randomized controlled trials: organized mammographic screening substantially reduces breast carcinoma mortality. *Cancer*. 2001;91(9):1724-1731.
- 9. The Swedish Organized Service Screening Evaluation Group. Reduction in breast cancer mortality from organized service screening with mammography: 1. Further confirmation with extended data. *Cancer Epidemiol*. 2006;15(1):45-51.
- 10. Coldman A, Phillips N, Wilson C, et al. Pan-Canadian Study of Mammography Screening and Mortality. Journal of the National Cancer Institute. Oct 2014;106(11):1-7.
- 11. Hofvind S, Ursin G, Tretli S, Sebuødegård S, Møller B. Breast cancer mortality in participants of the Norwegian Breast Cancer Screening Program. *Cancer*. Sep 2013;119(17):3106-3112.
- 12. Whelehan P, Evans A, Wells M, Macgillivray S. The effect of mammography pain on repeat participation in breast cancer screening: a systematic review. *Breast.* Aug 2013;22(4):389-394.
- 13. Dullum JR, Lewis EC, Mayer JA. Rates and correlates of discomfort associated with mammography. *Radiology*. Feb 2000;214(2):547-552.
- 14. Gupta R, Nayak M, Khoursheed M, Roy S, Behbehani Al. Pain during mammography: impact of breast pathologies and demographic factors. *Medical principles and practice*. Jul-Sep 2003;12(3):180-183.

GE Healthcare - Confidential

GE MWS DOC1991348 Ver: 1.0; 22/May/2017


Study No: 124.03-2017-GES-0002



- 15. Poulos A, Rickard M. Compression in mammography and the perception of discomfort. *Australasian Radiology*. Aug 1997;41(3):247-252.
- 16. Kornguth PJ, Rimer BK, Conaway MR, et al. Impact of patient-controlled compression on the mammography experience. *Radiology*. Jan 1993;186(1):99-102.
- 17. de Groot JE, Broeders MJ, Brandenhorst W, den Heeten GJ, Grimbergen CA. Mammographic compression after breast conserving therapy: controlling pressure instead of force. *Medical Physics*. Feb 2014;41(2).
- 18. de Groot JE, Branderhorst W, Grimbergen CA, den Heeten GJ, Broeders MJM. Towards personalized compression in mammography: A comparison study between pressure- and force-standardization. *Euorpean Journal of Radiology.* Mar 2015;84(3):384-391.
- 19. Sechopoulos I, Suryanarayanan S, Vedantham S, D'Orsi C, Karellas A. Radiation Dose to Organs and Tissues from Mammography: Monte Carlo and Phantom Study. *Radiology*. 2008;246:434-443.



### APPENDIX A - STUDY SCHEDULE

Table A.1 - Schedule of Study Procedures

| | Subject Visits* | | |
|---|---|---|---|
| Evaluation | Screening & Enrollment** | Visit 1** | Post Image Acquisition |
| Written Informed Consent | X | | |
| Patient Demographics | X | | |
| Inclusion criteria | X | | |
| Exclusion criteria | X | | |
| FFDM Exam, including patient-assisted compression for the breast of interest | | × | |
| Image acquisition data collection | | Х | |
| Image attribute review | | | X |

<sup>\*</sup>Subjects will be followed for AE reporting purposes from the time when they enter the imaging exam room until the time when they leave the imaging exam room at each visit. There will be no follow-up.

<sup>\*\*</sup> Screening, enrollment, and procedures may be conducted on the same day for study subjects.

**Study No:** 124.03-2017-GES-0002



### APPENDIX B - STUDY SITE AND INVESTIGATOR LIST

The following investigators at each study site will be responsible for the conduct of this study:

| Investigator(s):1 | Kathy Schilling, MD, Principal<br>Investigator | Boca Raton Regional Hospital Christine E. Lynn Women's Health and |
|---|---|---|
| | Tel: 1-561-955-5000 | Wellness Institute |
| | e-mail: kschilling@brrh.com | Address: 690 Meadows Road |
| | | Boca Raton, FL, 33486 U.S. |

<sup>&</sup>lt;sup>1</sup> The role of the *Principal Investigator* is to implement and manage the conduct of the investigation as well as ensure data integrity and the rights, safety, and well-being of humans involved in the study [ISO 14155:2011 9.1]. *Co-Investigators* share all responsibilities of the *Principal Investigator*, and *Sub-investigators* share only those responsibilities designated by the *Principal Investigator*.